CLINICAL TRIAL: NCT03245970
Title: Use of Impedance Cardiography to Decrease the Risk of Preeclampsia
Brief Title: Impedance Cardiography to Decrease the Risk of Preeclampsia
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Investigator retired. Other investigators did not want to continue study.
Sponsor: University of Tennessee Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4222
Record Dates: First submitted 2017-08-08; First posted 2017-08-10 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Chronic Hypertension Complicating Pregnancy (Diagnosis); Preeclampsia
MeSH Terms: conditions — Disease; Pre-Eclampsia | interventions — Labetalol; Nifedipine; Atenolol

STUDY DESIGN:
Intervention Model Description: Randomization to treatment or non treatment group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment Arm (Active Comparator): Treatment arm patients will be randomized to treatment with antihypertensive medications used with pregnancy for thirty years.
  Intervention: Labetalol Hydrocholoride 200 mg orally every 12 hours Nifedipine 60 mg orally daily Atenolol 25 mg daily
  Interventions: Drug: Labetalol Hydrocholoride 200 mg orally every 12 hours; Drug: Nifedipine 60 mg orally daily; Drug: Atenolol 25 mg daily
- Non Treatment (No Intervention): Non treatment Arm patients who are randomized to the non-treatment arm will not receive antihypertensive medications.

INTERVENTIONS:
Drug: Labetalol Hydrocholoride 200 mg orally every 12 hours — Anti-hypertensive prescribed for increased cardiac output as determined by impedance cardiography
  Other Names: Trandate
  Arms: Treatment Arm
Drug: Nifedipine 60 mg orally daily — Anti-hypertensive medication prescribed for increased systemic vascular resistance as determined by impedance cardiography
  Other Names: Procardia
  Arms: Treatment Arm
Drug: Atenolol 25 mg daily — Anti-hypertensive prescribed for increased cardiac output with tachycardia or maternal pulse rate 110 or greater
  Other Names: Tenormin
  Arms: Treatment Arm

SUMMARY:
To determine if the use of impedance cardiography can identify appropriate medications for use in treating chronic hypertensive patients to decrease the risk of preeclampsia.

DETAILED DESCRIPTION:
Impedance cardiography helps determine whether vasoconstriction or an elevated cardiac output is occurring. The test is easy to perform and non invasive. The treatment for an elevated cardiac output in pregnancy is a beta-blocker while a vasodilator is used for vasoconstriction. If a beta-blocker is given to someone that vasoconstricted, this might make the cardiovascular parameters worse, leading to no improvement in future pregnancy issues. Likewise, if a vasoconstricting drug is given to someone with an elevated cardiac output, it could potentially make the cardiovascular parameters worse.

All centers in the United States that choose to prescribe an antihypertensive medication for use in pregnancy do so by trial and error, whereas impedance cardiography can help the clinician choose the best medication from the start. Many pregnant patient patients have chronic hypertension and this population is at increased risk for superimposed preeclampsia and other pregnancy complications. The current recommendation for pregnancy is to NOT treat mild hypertension because studies have not shown any benefit. These studies, have also not shown any harm. Prior studies that have shown no benefit to treatment of mild hypertension in pregnancy may be hampered by choosing the wrong antihypertensive medication, thereby not improving the rate of superimposed preeclampsia and other pregnancy related complications.

ELIGIBILITY:
Inclusion Criteria:

Pregnant patients 18-51 years old Less than 20 weeks gestation with mild chronic hypertension - Not on antihypertensive medications

Exclusion Criteria:

Patients with an allergy to antihypertensive medication or contraindication for their usage such as certain cardiac or neurologic disorder during pregnancy Patients who have a blood pressure 140/90 or greater -

Ages: 18 Years to 51 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Rates of preeclampsia in chronically hypertensive pregnant women | 2 years
  Rates of preeclampsia in chronically hypertensive pregnant women

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Fortner, MD, Principal Investigator — University of Tennessee Medical Center
Locations (1):
- HIgh Risk Obstetrical Consultants, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No